CLINICAL TRIAL: NCT05240911
Title: Compare a New Method to the Traditional One to Estimate Levothyroxine Dose for Patients Needing Replacement Therapy After Total or Completion Thyroidectomy
Brief Title: Individual Dosing of Levothyroxine After Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-041
Record Dates: First submitted 2022-02-06; First posted 2022-02-15 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-01

CONDITIONS: Thyroid Neoplasms; Hypothyroidism; Surgery
Keywords: levothyroxine; thyroidectomy; thyroid hormone replacement therapy; individualized therapy; regression model
MeSH Terms: conditions — Thyroid Neoplasms; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poisson regression model dosing scheme (Experimental): daily levothyroxine dose=e[2.02+0.01(W)-0.0037(A )-0.098(F)-0.01(B)+0.007(T)+0.108(I)-0.014(M), where W is the weight of the patient (Kg), A is the age of the patient (years), and F is the gender (for women 1, male is 0), B represents the patient's body mass index (BMI), T represents the preoperative TSH level, I represents whether the patient takes iron preparations (1, if not 0), M represents whether the patient takes multivitamins/minerals (1, if not 0).
  Interventions: Drug: Levothyroxine Sodium Tablets
- weight-based dosing scheme (Active Comparator): daily levothyroxine dose=1.6 μg /kg/d
  Interventions: Drug: Levothyroxine Sodium Tablets

INTERVENTIONS:
Drug: Levothyroxine Sodium Tablets — For patients in experimental group, initial levothyroxine dose is calculated through the Poisson regression model; and for patients in comparator group, initial levothyroxine dose is calculated through 1.6 ug/kg/d.
  Other Names: LT4

SUMMARY:
Recently, Zaborek et al. raised a Poisson regression model for levothyroxine(LT4) dosing scheme to predict individual dose of LT4 after thyroidectomy: daily LT4 dose=e[2.02+0.01(W)-0.0037(A )-0.098(F)-0.01(B)+0.007(T)+0.108(I)-0.014(M), where W is the weight of the patient (Kg), A is the age of the patient (years), and F is the gender (for women 1, male is 0), B represents the patient's body mass index (BMI), T represents the preoperative TSH level, I represents whether the patient takes iron preparations (1, if not 0), M represents whether the patient takes multivitamins/minerals (1, if not 0). We demonstrated its value with our retrospective data in our center. Therefore, we intend to carry out this randomized controlled trial in order to further evaluate the model. The clinical significance of this method can provide a basis for the future use in clinical optimization of individualized dosing.

DETAILED DESCRIPTION:
Patients who underwent total/near-total thyroidectomy or completion thyroidectomy and require levothyroxine replacement therapy will be enrolled in this study. They will be randomized distributed into two groups. In one group, patients will be dosing LT4 according to weight-based algorithm, namely 1.6 μg /kg/d. In the other group, patients will be dosing LT4 according to the Poisson regression model algorithm. They will be followed up 3-6 weeks after surgery for the first time. During the follow up, thyroid hormone will be tested and LT4 dosing will be adjusted accordingly. Then, we compare patients in which group will achieve euthyroidism more quickly.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent total/near-total thyroidectomy or completion thyroidectomy; patients with benign disease, or low-risk differentiated thyroid cancer, or medullary thyroid cancer who don't need TSH suppressive therapy;

Exclusion Criteria:

* patients with heart disease or severe liver/kidney insufficiency; patients taking liothyronine in addition to levothyroxine;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
euthyroidism | 1 year
  a serum thyroid-stimulating hormone (TSH) level of 0.45 - 4.50 mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Qunzi Zhao, M.D., Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaborek NA, Cheng A, Imbus JR, Long KL, Pitt SC, Sippel RS, Schneider DF. The optimal dosing scheme for levothyroxine after thyroidectomy: A comprehensive comparison and evaluation. Surgery. 2019 Jan;165(1):92-98. doi: 10.1016/j.surg.2018.04.097. Epub 2018 Nov 6. PMID 30413325